CLINICAL TRIAL: NCT01189292
Title: Preoperative Single-dose Steroid Application for the Treatment of Nausea and Vomiting After Thyroid Surgery
Acronym: tPONV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Ignazio Tarantino, M.D:, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EKSG 10/082/2B
Record Dates: First submitted 2010-07-19; First posted 2010-08-26 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Thyroidectomy; Thyroid Diseases
Keywords: postoperative nausea and vomitus; PONV; thyroid surgery
MeSH Terms: conditions — Thyroid Diseases; Postoperative Nausea and Vomiting; Vomiting | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone injection (Active Comparator): Administration of 8mg(2ml) intravenous Dexamethasone (Mephameson®)
  Interventions: Drug: Dexamethasone
- Placebo (NaCl 0.9%) (Placebo Comparator)
  Interventions: Other: NaCl 0.9%

INTERVENTIONS:
Drug: Dexamethasone — 8mg (2ml) of dexamethasone (Mephameson®) administered intravenously preoperatively before thyroid surgery
  Other Names: Mephameson
  Arms: Dexamethasone injection
Other: NaCl 0.9% — 2ml of NaCl 0.9% administered intravenously preoperatively before thyroid surgery
  Arms: Placebo (NaCl 0.9%)

SUMMARY:
The study is to compare the postoperative recovery, as determined by postoperative nausea and vomiting (PONV) after preoperative application of single-dose dexamethasone versus saline in patients undergoing partial or total thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Planned partial or total thyroidectomy

Exclusion Criteria:

* History of adverse effects to dexamethasone or propyleneglycol or di-natrium-EDTA
* Patients with chronic pain
* Necessity for opioids-application in the postoperative course
* Not possible administration of a cervical block (0.5% bupivacaine at a dose of 20ml)
* Patients with Diabetes mellitus
* Pregnancy (test in young women)
* Glaucoma
* Patients who received antiemetic therapy within 48h before surgery
* Patients with acute pain requiring painkillers others than paracetamol or more than single dose NSAR treatment within 48h before surgery
* Use of psychotropic drugs
* Incompliant patients
* Preoperatively high suspicion of malignancy
* Re-operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clerici, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of Surgery, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] Tarantino I, Warschkow R, Beutner U, Kolb W, Luthi A, Luthi C, Schmied BM, Clerici T. Efficacy of a Single Preoperative Dexamethasone Dose to Prevent Nausea and Vomiting After Thyroidectomy (the tPONV Study): A Randomized, Double-blind, Placebo-controlled Clinical Trial. Ann Surg. 2015 Dec;262(6):934-40. doi: 10.1097/SLA.0000000000001112. PMID 25563879
- [Derived] Tarantino I, Beutner U, Kolb W, Muller SA, Luthi C, Luthi A, Schmied BM, Clerici T, Warschkow R. Study protocol for a randomized, double-blind, placebo-controlled trial of a single preoperative steroid dose to prevent nausea and vomiting after thyroidectomy: the tPONV study. BMC Anesthesiol. 2013 Sep 9;13(1):19. doi: 10.1186/1471-2253-13-19. PMID 24015953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients older than 18 years scheduled for a primary partial or total thyroidectomy due to benign disease at the Kantonsspital St. Gallen, Department of Surgery were recruited.
Period: Intention to Treat Analysis
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Started | 76 | 76
Completed | 76 | 76
Not Completed | 0 | 0
Period: Per Protocol Analysis
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Started | 76 | 76
Completed | 65 | 60
Not Completed | 11 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%) | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 67 | 137
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.0) | 48.4 (13.4) | 49.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 58 | 120
  Male | 14 | 18 | 32
Region of Enrollment [Number; unit: participants]
  Switzerland | 76 | 76 | 152
Body mass index [Mean (Standard Deviation); unit: kg/m²] | 24.8 (4.1) | 25.4 (4.6) | 25.1 (4.4)
Diagnosis [Number; unit: participants]
  Graves disease | 13 | 12 | 25
  Goiter, multinodular | 35 | 33 | 68
  Goiter, uninodular | 28 | 31 | 59
Type of surgery [Number; unit: participants]
  Hemithyroidectomy | 37 | 38 | 75
  Near total thyroidectomy | 19 | 13 | 32
  Total thyroidectomy | 20 | 25 | 45
Lymph node dissection (C1/level VI) [Number; unit: participants]
  no | 63 | 65 | 128
  yes | 13 | 11 | 24
Operating time [Mean (Standard Deviation); unit: minutes] | 126.2 (40.9) | 127.5 (45.7) | 126.8 (43.2)
Specimen weight [Mean (Standard Deviation); unit: gram] | 45.3 (40.1) | 51.2 (58.2) | 48.3 (49.9)
Histology of specimen [Number; unit: participants]
  Papillary thyroid cancer (PTC) | 3 | 7 | 10
  Follicular thyroid cancer (FTC) | 4 | 2 | 6
  Benign disease | 69 | 67 | 136

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Nausea and Vomiting
Description: Compare the postoperative recovery, as determined by postoperative nausea and vomiting (PONV) after preoperative application of single-dose dexamethasone versus saline in patients undergoing partial or total thyroidectomy (primary end-point)
  * any PONV event within 48 hours after surgery
  * PONV was measured at 4, 8, 16, 24, 32 and 48 hours after surgery
Time Frame: within 48 hours after surgery
Population: intention to treat analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Number analyzed (Participants) | 76 | 76
percentage of participants | 29 [20 to 40] | 57 [45 to 67]
Statistical Analysis 1: Comparison: Dexamethasone Injection vs Placebo (NaCl 0.9%); null hypothesis: Incidence of PONV is the same in both treatment arms; Test type: Superiority or Other; p = 0.001, Chi-squared; Risk Difference (RD) = 28, 95% CI 2-sided [12 to 42]

2. Secondary Outcome: Incidence of Postoperative Nausea and Vomiting
Description: as for outcome 1
Time Frame: within 48 hours after surgery (PP)
Population: per protocol analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Number analyzed (Participants) | 65 | 60
percentage of participants | 28 [18 to 40] | 52 [39 to 64]
Statistical Analysis 1: Comparison: Dexamethasone Injection vs Placebo (NaCl 0.9%); per protocol analysis; Test type: Superiority or Other; p = 0.006, Chi-squared; Risk Difference (RD) = 24, 95% CI 2-sided [7 to 40]

3. Secondary Outcome: Degree of Post Operative Nausea and Vomiting
Description: mild nausea:......single administration of an antiemetic drug
  severe nausea: repeated administration of antiemetic drugs
  vomiting:...........at least one vomiting event
Time Frame: 4 hours after surgery
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Number analyzed (Participants) | 76 | 76
participants
  mild nausea | 9 | 15
  severe nausea | 1 | 3
  vomiting | 3 | 12

4. Secondary Outcome: Degree of Post Operative Nausea and Vomiting
Description: as for outcome 3
Time Frame: 8 hours after surgery
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Number analyzed (Participants) | 76 | 76
participants
  mild nausea | 5 | 7
  severe nausea | 0 | 3
  vomiting | 8 | 12

5. Secondary Outcome: Postoperative Pain After Physical Stress
Description: Compare grade of pain between the treatment (dexamethasone) and the control (saline) group
  * Pain was measured using a verbal rating scale ranging from 0 (no pain) to 10 in steps of 1
  * before obtaining the pain rating, patients were asked to turn their heads (physical stress)
Time Frame: 4 and 8 hours after surgery
Population: intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Number analyzed (Participants) | 76 | 76
units on a scale
  4 hours after surgery | 1.88 (1.52) | 2.09 (1.73)
  8 hours after surgery | 1.88 (1.54) | 2.01 (1.75)
Statistical Analysis 1: Comparison: Dexamethasone Injection vs Placebo (NaCl 0.9%); Test type: Superiority or Other; p = 0.674, Mixed Models Analysis; mixed model over the mean ranks at all time points measured (4, 8, 16, 24, 32, 48 hours)

6. Secondary Outcome: Length of Hospital Stay
Description: Compare the lengths of hospital stay between the treatment (dexamethasone) and the control (saline) group
Time Frame: Difference between day of admission and day of discharge
Population: intention to treat
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Number analyzed (Participants) | 76 | 76
hour | 48.3 (15.7) | 48.1 (12.6)
Statistical Analysis 1: Comparison: Dexamethasone Injection vs Placebo (NaCl 0.9%); Test type: Superiority or Other; p = 0.835, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Necessary Anesthesiological Medication
Description: Compare the amount of necessary anesthesiologic medication during the operation between the treatment (dexamethasone) and the control (saline) group
Time Frame: measured from beginning of anaesthesia to end of anaesthesia
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Number analyzed (Participants) | 76 | 76
milligram
  Propofol | 1097 (422) | 1168 (422)
  Remifentanil | 1.944 (1.197) | 1.978 (1.111)
  Fentanyl | 0.427 (0.111) | 0.444 (0.108)
  Rocuronium | 38.7 (7.3) | 39.7 (8.3)

ADVERSE EVENTS:
Time Frame: during hospitalisation (on average 2 days)
Description: adverse events were recorded during the hospital stay
Arm/Group | Dexamethasone Injection | Placebo (NaCl 0.9%)
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 8/76 | 9/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Injection (N=76) | Placebo (NaCl 0.9%) (N=76)
surgical adverse event grade I (Surgical and medical procedures) | 4 | 2 — for example: recurrent laryngeal nerve palsy, hoarseness, minor bleeding
temporary hypoparathyroidism (Endocrine disorders) | 2 | 2 — Grade 2 on Clavien-Dindo scale
bleeding requiring reoperation (Surgical and medical procedures) | 1 | 0
medical adverse events grade 1 (General disorders) | 1 | 2 — for example: coughing, sinus tachycardia, temporary compensated renal insufficiency
Allergic reaction to metamizole (Immune system disorders) | 0 | 1 — CTCAE grade 2
hypocalcemia (Endocrine disorders) | 0 | 2 — CTCAE grade 2

LIMITATIONS AND CAVEATS:
all patients received a bilateral superficial cervical plexus block during surgery which could explain the very low postoperative pain scores compared to other similar studies

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes